CLINICAL TRIAL: NCT05417646
Title: Impact of SGLT2 on Glucosuria in HNF1A-MODY
Acronym: MOD3ST-CLAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-21066984
Record Dates: First submitted 2022-05-24; First posted 2022-06-14 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Maturity-Onset Diabetes of the Young, Type 3; Type 2 Diabetes
Keywords: Sodium-Glucose Transporter 2; Sodium-Glucose Transporter 2 Inhibitors; Glycosuria
MeSH Terms: conditions — Maturity-Onset Diabetes of the Young, Type 3; Diabetes Mellitus, Type 2; Glycosuria | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- HNF1A-MODY - SGLT2 inhibition (Active Comparator): 3-hour hyperglycemic clamp with inhibition of SGLT2 (single-dose empagliflozin 25 mg two hours before clamp)
  Interventions: Other: Hyperglycaemic clamp; Drug: Empagliflozin
- HNF1A-MODY - Placebo (Placebo Comparator): 3-hour hyperglycemic clamp without inhibition of SGLT2 (placebo comparator to empagliflozin)
  Interventions: Other: Hyperglycaemic clamp; Drug: Placebo
- Type 2 Diabetes - SGLT2 inhibition (Active Comparator): 3-hour hyperglycemic clamp with inhibition of SGLT2 (single-dose empagliflozin 25 mg two hours before clamp)
  Interventions: Other: Hyperglycaemic clamp; Drug: Empagliflozin
- Type 2 Diabetes - Placebo (Placebo Comparator): 3-hour hyperglycemic clamp without inhibition of SGLT2 (placebo comparator to empagliflozin)
  Interventions: Other: Hyperglycaemic clamp; Drug: Placebo

INTERVENTIONS:
Other: Hyperglycaemic clamp — Three-hour, three-step glucose clamp with plasma glucose targets 10, 14 and 18 mmol/l (each one hour)
Drug: Placebo — Placebo comparator to empagliflozin
  Arms: HNF1A-MODY - Placebo; Type 2 Diabetes - Placebo
Drug: Empagliflozin — Single-dose, 25 mg, two hours before clamp
  Arms: HNF1A-MODY - SGLT2 inhibition; Type 2 Diabetes - SGLT2 inhibition

SUMMARY:
Maturity onset diabetes of the young (MODY) is a subtype of diabetes which is caused by mutations in specific genes leading to diabetes. The most common cause of MODY is due to mutations in the gene hepatocyte nuclear factor 1 alpha (HNF1A) and is consequently named HNF1A-MODY (or MODY3). HNF1A-MODY is associated with urinary excretion of glucose at lower blood glucose levels compared to other types of diabetes. Normally, glucose is reabsorbed by sodium-glucose cotransporter 2 (SGLT2), but SGLT2 is downregulated due to the mutation in HNF1A. Investigators aim to evaluate the impact of the decreased expression of SGLT2 on glucosuria in patients with HNF1A-MODY compared to patients with type 2 diabetes (T2D) using a single dose of an SGLT2 inhibitor during a glucose clamp experiment.

DETAILED DESCRIPTION:
Participants: Patients with HNF1A-MODY (n=12) and patients with T2D (n=12)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* HNF1A-MODY verified by genetic testing (only patients with HNF1A-MODY)
* Type 2 diabetes diagnosis according to World Health Organization (only patients with type 2 diabetes)
* Treatment with diet and/or a glucose-lowering drug (only patients with HNF1A-MODY)
* Normal haemoglobin (males 8.3-10.5 mmol/l, females 7.3-9.5 mmol/l)
* Informed consent

Exclusion Criteria:

* Nephropathy (estimated GFR <60 ml/min/1.73m2 and/or albuminuria)
* Known significant liver disease and/or plasma alanine aminotransferase (ALT) and/or plasma aspartate aminotransferase (AST) above 2 × normal values)
* Pregnancy or breastfeeding
* Treatment with SGLT2 inhibitor
* Fasting plasma glucose > 10 mmol/l
* Family history of HNF1A-MODY (only patients with type 2 diabetes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Urinary glucose excretion | Assesed during 3 hour hyperglycaemic clamp

SECONDARY OUTCOMES:
Urinary glucose excretion adjusted for glomerular filtration rate (GFR) | Assesed during 3 hour hyperglycaemic clamp
  GFR: 99mTc-diethylenetriaminepentaacetic acid (99mTc-DTPA) plasma clearance
Infused amount of glucose | Assesed during 3 hour hyperglycaemic clamp
Urine volume | Assesed during 3 hour hyperglycaemic clamp
Glucose tissue disposal | Assesed during 3 hour hyperglycaemic clamp
  difference between infused and excreted glucose
Urinary creatinine clearance | Assesed during 3 hour hyperglycaemic clamp
  Urinary creatinine clearance calculated by plasma creatinine concentration and urinary creatinine excretion
Concentration of plasma c-peptide | Assesed during 3 hour hyperglycaemic clamp
  Summarized as area under the curve (AUC)
Concentration of plasma glucagon | Assesed during 3 hour hyperglycaemic clamp
  Summarized as AUC
Renal threshold of glucose excretion | Assesed during 3 hour hyperglycaemic clamp
  Estimated using plasma glucose concentrations, urinary glucose excretion and GFR

CONTACTS AND LOCATIONS:
Overall Officials: Tina Vilsbøll, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No